CLINICAL TRIAL: NCT03684941
Title: Evaluation of a New Catheter Coating Process for Urinary Catheters Used for Intermittent Catheterization - A Prospective, Blinded, Randomized, Cross-over, Multicenter Study
Brief Title: Evaluation of a New Catheter Coating Process for Urinary Catheters Used for Intermittent Catheterization.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dentsply International (Industry)
Collaborators: Wellspect HealthCare (Industry)
Responsible Party: Sponsor
Organization: Dentsply Sirona Inc. (Industry)
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: LOF-0034
Record Dates: First submitted 2018-09-17; First posted 2018-09-26 (Actual); Last update posted 2018-12-05 (Actual); Status verified 2018-12

CONDITIONS: Intermittent Urethral Catheterization

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Treatment Period One (Experimental): LoFric, hydrophilic urinary catheter for single use. The study device is based on commercially available hydrophilic urinary catheters for intermittent catheterization, but with a different coating process than the comparator. Treatment Period One will last 1 week.
  Interventions: Device: Treatment Period One
- Treatment Period Two (Active Comparator): CE-marked LoFric®, hydrophilic urinary catheter for single use. The comparator product is today commercially available and produced by WHC. Treatment Period Two will last 1 week.
  Interventions: Device: Treatment Period Two

INTERVENTIONS:
Device: Treatment Period One — LoFric Origo urinary catheter, 40-cm length, CH12/CH14 diameter, with Nelaton tip
  Arms: Treatment Period One
Device: Treatment Period Two — CE-marked LoFric Origo urinary catheter, 40-cm length, CH12/CH14 diameter, with Nelaton tip
  Arms: Treatment Period Two

SUMMARY:
This is a prospective, double-blinded, randomized, multi-centre, cross-over study. All subjects will use both the study device (test catheter) and the comparator (control catheter) for one week each.

ELIGIBILITY:
Inclusion Criteria:

* Provision of informed consent.
* Males, aged 18 years and over.
* Maintained urethra sensibility as judged by the subject. (Can you feel the catheter during catheterization? Yes.).
* Practice CIC at least 2 times daily.
* Using catheters in the size CH 12 or CH 14, Nelaton tip, and able to use catheter length of 40 cm.
* Experienced users of CIC defined as a minimum of three months on therapy.
* Adults able to read, write and understand information given to them regarding the study.

Exclusion Criteria:

* Ongoing, symptomatic UTI at enrolment as judged by investigator. The definition of UTI, is a positive urine culture of ≥103 CFU/ml of ≥1 bacterial species and presence of symptoms or signs compatible with UTI with no other identified source of infection.
* Known urethral stricture which, in the opinion of the investigator, could influence the subject's evaluation of the catheters.
* Involvement in the planning and conduct of the study (applies to both WHC staff and staff at the study site).
* Previous enrolment or randomisation of treatment in the present study.
* Simultaneous participation in another clinical study that may impact the primary endpoint.
* Severe non-compliance to protocol as judged by the investigator

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2018-08-29 (Actual); Primary Completion 2018-11-19 (Actual); Study Completion 2018-11-19 (Actual)

PRIMARY OUTCOMES:
Tolerability of practicing CIC by using two urinary catheters produced with different coating processes measuring change over time by means of subjective assessment scales | 2 weeks in total. 1 week Treatment Period One/1 week Treatment Period Two
  The primary objective of this study is to compare the subjects' tolerability of practising CIC by using two urinary catheters produced with different coating processes by means of subjective assessment scales.

SECONDARY OUTCOMES:
Tolerability with regards to perceived pain, when using two different urinary catheters; test vs control catheter. | 2 weeks in total. 1 week Treatment Period One/1 week Treatment Period Two. Safety variables spontaneously reported during whole study period
  AE/SAE/ADE/SADE reporting/PRO variables. Assessed in patient questionnaire for each subject. A 5 graded scale will be used to determine the perception and the severity of each variable. The difference between the treatments will be calculated for each subject.
Tolerability with regards to presence of bleeding, when using two different urinary catheters; test vs control catheter | 2 weeks in total. 1 week Treatment Period One/1 week Treatment Period Two. Safety variables spontaneously reported during whole study period
  AE/SAE/ADE/SADE reporting /PRO variables. Assessed in patient questionnaire for each subject. A 5 graded scale will be used to determine the perception and the severity of each variable. The difference between the treatments will be calculated for each subject.
Tolerability with regards to perceived "other discomfort", when using two different urinary catheters; test vs. control catheter | 2 weeks in total. 1 week Treatment Period One/1 week Treatment Period Two. Safety variables spontaneously reported during whole study period
  PRO variables. Frequency of "other discomfort" (yes/ no) will be assessed in patient questionnaire. The frequency of "other discomfort" will be compared between the treatments. "Other discomfort" will be further specified using 5 graded scale (as for the other variables on the 5 graded scale the difference between the treatments will be calculated for each subject).
Perception of the catheter's slipperiness, smoothness, flexibility, usability, and resistance, when practicing intermittent self-catheterization with urinary catheters; test vs. control catheter | 2 weeks in total. 1 week Treatment Period One/1 week Treatment Period Two. Safety variables spontaneously reported during whole study period
  PRO variables. Assessed in patient questionnaire for each subject. A 5 graded scale will be used to determine the perception and the severity of each variable. The difference between the treatments will be calculated for each subject.
To evaluate subject satisfaction with catheter; test vs. control catheter. | 2 weeks in total. 1 week Treatment Period One/1 week Treatment Period Two. Safety variables spontaneously reported during whole study period
  PRO variables. Assessed in patient questionnaire for each subject. A 5 graded scale will be used to determine the satisfaction. The difference between the treatments will be calculated for each subject.
Total number of DD/AE/SAE/ADE/SADE/ USADE. | 2 weeks in total.
  Total number of DD/AE/SAE/ADE/SADE/ USADE observed by the study personnel or spontaneously reported from subject will be calculated. The frequency of DD/AE/SAE/ADE/SADE/ USADE will be calculated for each treatment group.

CONTACTS AND LOCATIONS:
Locations (8):
- Sweden (8):
  - Urologcentrum Borås, Borås
  - Urologkliniken vid Carlanderska AB, Gothenburg
  - Specialistmottagningen i Urologi, Halmstad, Halmstad
  - Urologmottagningen, Centralsjukhuset Karlstad, Karlstad
  - Urologiska kliniken, Urologmottagningen Universitetssjukhuset Örebro, Örebro
  - GHP Urologcentrum Stockholm, Stockholm
  - Uroterapimottagningen, Sjukhuset Torsby, Torsby
  - Urologmottagningen, Akademiska sjukhuset, Uppsala